CLINICAL TRIAL: NCT04688879
Title: Thrombolysis With Intra-arterial Urokinase for Acute Superior Mesenteric Artery Occlusion: Outcome Analysis
Brief Title: Thrombolysis With Intra-arterial Urokinase
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Being-Chuan Lin, Attending doctor of the Trauma & Emergency Surgery, Chang Gung Memorial Hospital
Other Study IDs: 202000381B0
Record Dates: First submitted 2020-12-27; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Arterial Occlusion Mesenteric Artery Superior
Keywords: intra-arterial urokinase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- According to the degree of occlusion, 13 patients were divided into complete and incomplete groups.: Seven patients were complete occlusion and 6 patients were incomplete occlusion and all underwent thrombolysis with intra-arterial urokinase and the outcome was analysed..
  Interventions: Procedure: intra-arterial urokinase thrombolysis

INTERVENTIONS:
Procedure: intra-arterial urokinase thrombolysis — Under local anaesthesia, the right femoral artery was punctured in accordance with the Seldinger technique, and a 6-Fr sheath, 10 cm in length, was implanted. Selective catheterization of the SMA was performed with 4-Fr catheter. The SMA angiography was performed to identify the filling defect. Thrombolysis was performed using a 5-Fr multiple-sideport infusion catheter (100cm with sideport of 7cm, 14 ports or 100cm with sideport of 15cm, 30 ports, Cook, Bloomington, IN, U.S.A). The tip of the microcatheter was embedded in the thromboembolism, which was fragmented at the time of thrombolysis. Thrombolysis was performed locally in the SMA with a bolus of urokinase

SUMMARY:
Patients with acute superior mesenteric artery (SMA) occlusion were included in this study. The clinical presentation and effect of the recanalization of the SMA was analyzed on follow-up angiography.

DETAILED DESCRIPTION:
Thirteen patients with acute SMA occlusion who underwent intra-arterial urokinase thrombolysis between 2008 and 2020 were retrospectively evaluated.

Clinically, the abdominal pain and the effect of the SMA on angiography will be compared in response and non-response groups.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of SMA occlusion

Exclusion Criteria:

* shock in the triage screening
* peritonitis
* 3. intramural gas, mesenteric or portal venous gas on contrast-enhanced abdominal CT

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 13
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Thrombolysis with intra-arterial urokinase for acute superior mesenteric artery occlusion: Outcome analysis | Daily series follow-up angiography in the next 72 hours after thrombolysis with intra-arterial urokinase.
  Degree of patency and appearance of the SMA will be analyzed in the follow-up angiography.

CONTACTS AND LOCATIONS:
Overall Officials: Being-Chuan Lin, Study Director — Chang Gung Hospital
Locations (1):
- Chang Gung memorial Hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bala M, Kashuk J, Moore EE, Kluger Y, Biffl W, Gomes CA, Ben-Ishay O, Rubinstein C, Balogh ZJ, Civil I, Coccolini F, Leppaniemi A, Peitzman A, Ansaloni L, Sugrue M, Sartelli M, Di Saverio S, Fraga GP, Catena F. Acute mesenteric ischemia: guidelines of the World Society of Emergency Surgery. World J Emerg Surg. 2017 Aug 7;12:38. doi: 10.1186/s13017-017-0150-5. eCollection 2017. PMID 28794797
- [Result] Bjornsson S, Bjorck M, Block T, Resch T, Acosta S. Thrombolysis for acute occlusion of the superior mesenteric artery. J Vasc Surg. 2011 Dec;54(6):1734-42. doi: 10.1016/j.jvs.2011.07.054. Epub 2011 Sep 1. PMID 21889287
- [Result] Tilsed JV, Casamassima A, Kurihara H, Mariani D, Martinez I, Pereira J, Ponchietti L, Shamiyeh A, Al-Ayoubi F, Barco LA, Ceolin M, D'Almeida AJ, Hilario S, Olavarria AL, Ozmen MM, Pinheiro LF, Poeze M, Triantos G, Fuentes FT, Sierra SU, Soreide K, Yanar H. ESTES guidelines: acute mesenteric ischaemia. Eur J Trauma Emerg Surg. 2016 Apr;42(2):253-70. doi: 10.1007/s00068-016-0634-0. PMID 26820988